CLINICAL TRIAL: NCT04944043
Title: A Single Group, Open-Label, Multicenter ,Phase Ib/II Clinical Trials of TQ05105 Tablet in Patients With Glucocorticoid Refractory and Dependent Moderate to Severe Chronic Graft Versus Host Disease (cGVHD).
Brief Title: A Study of TQ05105 in Patients With Chronic Graft Versus Host Disease
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Chia Tai Tianqing Pharmaceutical Group Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: TQ05105-Ib/II-02
Record Dates: First submitted 2021-06-21; First posted 2021-06-29 (Actual); Last update posted 2025-12-03 (Actual); Status verified 2025-12

CONDITIONS: Chronic Graft Versus Host Disease
MeSH Terms: conditions — Bronchiolitis Obliterans Syndrome

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TQ05105 Tablet (Experimental): TQ05105 tablet 10mg given orally, twice daily in 28-cycle.
  Interventions: Drug: TQ05105 Tablet

INTERVENTIONS:
Drug: TQ05105 Tablet — TQ05105 tablet is a Janus Kinase (JAK) inhibitor, which can inhibit the abnormal activation of JAK 2-V617F mutation, thereby inhibiting the sustained abnormal activation of JAK / STAT pathway.

SUMMARY:
This study was a single arm, open label, multicenter phase Ib / II trial in subjects with glucocorticoid refractory / dependent moderate to severe cGVHD.The trial consisted of two phases: phase I for the dose exploration and phase II for the extension study.

ELIGIBILITY:
Inclusion Criteria:

* Understood and signed an informed consent form.
* ≥18 years old, Karnofsky Performance Scale of ≥60, life expectancy ≥ 6 months.
* Has received allogeneic hematopoietic stem cell transplantation (alloSCT).
* Clinically diagnosed moderate to severe cGVHD according to NIH Consensus Criteria.
* Has received systemic or topical corticosteroids therapy and confirmed steroid-refractory/dependent cGVHD according to NIH Consensus Criteria.
* Has received at least 1 lines of therapy for cGVHD.
* Adequate laboratory indicators.
* No pregnant or breastfeeding women, and a negative pregnancy test.

Exclusion Criteria:

* Has active acute GVHD.
* Has previously failed to respond to JAK inhibitors for GVHD, or who had used JAK inhibitors within 4 weeks before the first administration.
* Has uncontrollable active infections or infections requiring systematic treatment within 7 days before the first administration.
* Development of other basic diseases.
* Has malignant tumors within 3 years.
* Has multiple factors affecting oral medication.
* Has substance abuse or a psychotic disorder.
* Has severe and / or uncontrolled disease.
* Allergic to drugs or its constituents.
* Has participated in any other clinical trials within 4 weeks before first administration.
* According to the judgement of the investigators, there are other factors that may lead to the termination of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2021-06-25 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Maximal Tolerable Dose (MTD) | Baseline up to 4 weeks
  If dose limiting toxicity (DLT) occurs in 2 or more subjects in a given dose group, the dose level in the previous dose group is considered MTD. (Patients in phase Ib)
Recommended phase II dose (RP2D) | Baseline up to 4 weeks
  Recommended dose for phase II (Patients in phase Ib)
Best Overall Response Rate (BOR) | Baseline up to 96 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR). (Patients in phase II)

SECONDARY OUTCOMES:
Overall Response Rate (ORR) | Baseline up to 52 weeks
  Percentage of participants achieving complete response (CR) and partial response (PR) during the study according to the cGVHD NIH Consensus Criteria.
Duration of Response (DOR) | Baseline up to 96 weeks
  DOR defined as time from earliest date of disease response to earliest date of disease progression.
Overall survival (OS) | Baseline up to death event, up to 5 years.
  OS defined as the time from randomization to the time of death from any cause.
Non-relapse mortality (NRM) | Baseline up to 96 weeks
  Defined as the date of first dose to the date of death from non hematologic disease recurrence / progression
Failure Free Survival (FFS) | Baseline up to 12 months
  Defined as absence of relapse, death, or need for additional systemic immunosuppressant cGVHD therapy.
Changes in glucocorticoid dose | Baseline up to 96 weeks
  The reduction in glucocorticoid requirement would be regarded as an effect of the trial drug.
Changes in symptom burden | Baseline up to 96 weeks
  Evaluate changes in symptom burden as measured by the Lee Symptom Scale. A change of 7 points on the Lee Symptom Scale will be considered clinically significant and relates to improvement in quality of life.
Maximum plasma concentration (Cmax) | Pre-dose, 5, 15 , 30 minutes, 1 , 2 , 3 , 6, 8, 11 hours post-dose of day 1; Pre-dose of day 3,day5, day 6 ;Pre-dose, 5, 15 , 30 minutes, 1 , 2 , 3 , 6, 8, 11 hours post-dose of day 7.
  Cmax is the maximum plasma concentration of TQ05105 or its metabolite(s).
Time to reach maximum plasma concentration (Tmax) | Pre-dose, 5, 15 , 30 minutes, 1 , 2 , 3 , 6, 8, 11 hours post-dose of day 1; Pre-dose of day 3,day5, day 6 ;Pre-dose, 5, 15 , 30 minutes, 1 , 2 , 3 , 6, 8, 11 hours post-dose of day 7.
  To characterize the pharmacokinetics of TQ05105 by assessment of time to reach maximum plasma concentration.
Area under the plasma concentration time curve (AUC0-t) | Pre-dose, 5, 15 , 30 minutes, 1 , 2 , 3 , 6, 8, 11 hours post-dose of day 1; Pre-dose of day 3,day5, day 6 ;Pre-dose, 5, 15 , 30 minutes, 1 , 2 , 3 , 6, 8, 11 hours post-dose of day 7.
  To characterize the pharmacokinetics of TQ05105 by assessment of area under the plasma concentration time curve from zero to infinity.
Incidence rate of adverse event | Baseline up to 96 weeks.
  The occurrence rate of all adverse events (AEs), serious adverse events (SAEs) and treatment-related adverse events (TEAEs) assessed based on National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE) Version 5.0.

CONTACTS AND LOCATIONS:
Locations (12):
- China (12):
  - The First Affiliated Hospital of USTC (Anhui Provincial Hospital), Hefei, Anhui
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Nanfang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Guangzhou First People's Hospital, Guangzhou, Guangdong
  - The First Affiliated Hospital of Guangxi Medical University, Nanning, Guangxi
  - The Second Hospital of Hebei Medical University, Shijiazhuang, Hebei
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Union Hospital Tongji Medical College Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital Tongji Medical College of HUST, Wuhan, Hubei
  - The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu
  - Institute of Hematology & Blood Diseases Hospital, Chinese Academy of Medical Sciences & Peking Union Medical College, Tianjin, Tianjin Municipality
  - The First Affiliated Hospital, Zhejiang University School of Medicine, Hanzhou, Zhejiang

REFERENCES:
- [Derived] Zhao YM, Luo Y, Shi JM, Wang SQ, Wang CK, Jiang EL, Liang C, Zhu XY, Zhang XJ, Meng FK, Jin H, Zhao YQ, Yu J, Lai XY, Liu LZ, Fu HR, Ye YS, Zhang CX, Wang T, Tu LF, Wang XQ, Huang H. A first-in-class JAK/ROCK inhibitor, rovadicitinib, for glucocorticoid-refractory or -dependent chronic GVHD. Blood. 2025 Jun 12;145(24):2857-2872. doi: 10.1182/blood.2024026581. PMID 40009501